CLINICAL TRIAL: NCT02561507
Title: Use of Aspirin in the Perioperative Setting: A Surgeon's Survey
Brief Title: Perioperative Aspirin Usage Survey
Status: Terminated | Type: Observational
Why Stopped: This is not a clinical trial and was inadvertently entered into the system.
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Other Study IDs: 15-215
Record Dates: First submitted 2015-09-24; First posted 2015-09-28 (Estimated); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Surgery; Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- American College of Surgeons members: Survey participants
  Interventions: Behavioral: Survey

INTERVENTIONS:
Behavioral: Survey

SUMMARY:
This is a survey of members of the American College of Surgeons (ACS), to describe and explore current patterns of their decisions about withholding or continuation for patients taking aspirin (ASA) in the perioperative period. Secondarily, the survey will also explore surgeons' knowledge about the risks and benefits attending this decision, and about national organizations' recommendations.

DETAILED DESCRIPTION:
An announcement of the survey and invitation to participate will be posted in the "ACS Surgery News" newsletter published by the American College of Surgeons. Surgeons of all specialties will be invited to participate. No identifiers will be maintained with survey responses. In addition to the substantive questions below, typical demographic data will be obtained including participants' duration of practice, specialty, gender, state, etc.

The survey will include questions intended to characterize current practice surrounding the decision to continue or withhold aspirin in the perioperative period. Other questions will focus on surgeons' knowledge of national medical/surgical organizations that have published guidelines on the perioperative use of aspirin. Finally, other survey questions will characterize surgeons' knowledge of the platelet rebound effect.

ELIGIBILITY:
Inclusion Criteria:

* Members of the American College of Surgeons

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Members of the American College of Surgeons
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Typical proportion of participants' patients given a recommendation to stop taking aspirin | At time of survey; generally less than 20 minutes
Proportion of participants correctly identifying national organizations with perioperative aspirin recommendations | At time of survey; generally less than 20 minutes
Proportion of participants correctly answering questions about platelet rebound effect | At time of survey; generally less than 20 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Neal Gerstein, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico Hospital, Albuquerque, New Mexico, United States